CLINICAL TRIAL: NCT02056288
Title: A Randomized Comparison of Ultrasound Guided Supraclavicular Block(UGSB) and General Anesthesia (GA) to IV Narcotics and General Anesthesia for Postoperative Pain Relief in Children With Supracondylar Fractures.
Brief Title: A Comparison of UGSB and GA to IV Narcotics and GA for Post-Op Pain in Children With Supracondylar Fractures.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment was suspended due to the duration of the study and poor follow-up response by participants.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Chris Glover, Medical Director of Perioperative Services, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-27386
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Supracondylar Fractures
MeSH Terms: interventions — Fentanyl; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound Guided Supraclavicular block (Active Comparator): Patients randomized to the supraclavicular block group will receive an ultrasound guided nerve block with 0.2 ml/kg ropivacaine 0.5% (maximum 10 ml), using the technique described by Marhofer et al. In order to decrease variance in success rates, the ultrasound guided nerve block will be performed by 1 of the 4 anesthesiology co-investigators, each of whom have successfully performed over 100 ultrasound guided blocks in the past. Supraclavicular blocks were performed using the higher frequency of the probe and placing it in a coronal-oblique-plane in the supraclavicular fossa.
  Interventions: Drug: Ropivacaine
- IV Opioids (Active Comparator): Patients randomized to the systemic analgesia group will receive 1mcg/kg of fentanyl IV after induction.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Patients randomized to the systemic analgesia group will receive 1mcg/kg of fentanyl IV after induction.
  Arms: IV Opioids
Drug: Ropivacaine — Patients randomized to the systemic analgesia group will receive 1mcg/kg of fentanyl IV after induction. Patients randomized to the supraclavicular block group will receive an ultrasound guided nerve block with 0.2 ml/kg ropivacaine 0.5% (maximum 10 ml).
  Arms: Ultrasound Guided Supraclavicular block

SUMMARY:
This study compares nerve blocks to IV pain medicines in children with broken arms. We are trying to see if blocking the nerves in the broken arm results in better pain control and less side effects than injections of morphine into a vein after surgery for a broken elbow.

DETAILED DESCRIPTION:
Written consent will be obtained by the investigators prior to the surgical procedure using the Institutional Review Board (IRB) approved consent form. The medical record will be examined and the use of any analgesic medications in the 24 hours prior to the procedure will be recorded. Patients will be taken to the OR and anesthetized using standard procedures of the Texas Children's Hospital (TCH) department of anesthesia, including monitoring according to the American Society of Anesthesiologists guidelines (EKG, pulse oximetry, BP, temperature and end-tidal expired carbon dioxide and inhalation anesthetic gases). If the Attending Anesthesiologist believes the child is at risk for aspiration of gastric contents, a rapid sequence induction with propofol 3-4 mg/kg and succinylcholine 1mg/kg IV will be performed with cricoid pressure, in keeping with standard practices. In other patients an IV will be started after induction of anesthesia. An age appropriate endotracheal tube or appropriate sized laryngeal mask airway (LMA) will be inserted in all patients. Anesthesia will be maintained with sevoflurane, nitrous oxide and oxygen, adjusted to keep blood pressure and heart rate within 20% of baseline values, in keeping with standard practices. All patients will receive ketorolac 0.5mg/kg IV.

Patients will be randomized in a 1:1 ratio into one of two study groups: ultrasound guided supraclavicular block or IV opioids, based on a computer generated random number by using Random Allocation Software For Parallel Group Randomized Trials. The assignment will be made only after written informed consent has been obtained. There will be an equal chance a child will be assigned to one of the two groups. Patients randomized to the systemic analgesia group will receive 1mcg/kg of fentanyl IV after induction. Patients randomized to the supraclavicular block group will receive an ultrasound guided nerve block with 0.2 ml/kg ropivacaine 0.5% (maximum 10 ml), using the technique described by Marhofer et al. In order to decrease variance in success rates, the ultrasound guided nerve block will be performed by 1 of the 4 anesthesiology co-investigators, each of whom have successfully performed over 100 ultrasound guided blocks in the past. Supraclavicular blocks were performed using the higher frequency of the probe and placing it in a coronal-oblique-plane in the supraclavicular fossa. The brachial plexus will be identified as a cluster of hypoechoic nodules, lateral to the round pulsating hypoechoic subclavian artery and lying on top of the hyperechoic first rib. The cupola of the lung will be identified. If the transverse colli artery is visualized cephalically surrounding the plexus, the probe will be moved toward a better coronal oblique plane, directing the ultrasound beam slightly caudally, in order to keep the artery away from the plexus. The needle will be was carefully introduced using an in-plane (IP) technique from lateral to medial, toward but not into the brachial plexus. The entire needle image will be visualised at all times to ensure it does not enter the vessel, nerve plexus or pleura. The spread of local anesthetic to all targets of the plexus will be observed on the ultrasound image.

The time taken to place the block will be recorded from the time the ultrasound probe is first placed on the child until completion of local anesthetic injection. The observer collecting postoperative data will not be present when the block is placed, and a band-aid will be placed over the supraclavicular fossa in all patients to maintain blinding of the observer to the group assignment. During the operation patients can receive intraoperative fentanyl, 1 mcg/kg IV at a time, if the attending anesthesiologist believes it is clinically indicated. At the end of the operation, anesthetic gases will be discontinued while the patient breathes 100% oxygen. The trachea will be extubated when the patient responds to commands, and the child will then be taken to the Post Anesthetic Care Unit (PACU) in keeping with standard practices . A validated pain scale (verbal rating scale where 0 = no pain and 10 = worst possible pain ever) will be used throughout to assess the severity of pain in the postoperative period. In keeping with current practice, patients with pain scores>4 will be treated with morphine 0.05mg/kg IV at 10 minute intervals until the score is below 4. Oral acetaminophen with hydrocodone (Lortab elixir 0.15mg/kg hydrocodone) will be administered to children for pain scores between 2- 3. Supplemental oxygen, rescue antiemetic and antipruritic drugs will be administered in keeping with standard practices of TCH and the clinical judgment of the Attending Anesthesiologist. The duration of supplemental oxygen therapy, any medication administered and complications (side effects such as nausea, vomiting, itching, respiratory depression, prolonged awakening) will be recorded on the case report form.

The blinded observer will record pain scores within 15 minutes of arrival in the PACU and at 30 minutes, 1,2,6,12,24, and 48 hours after arrival in the PACU. If the child is sleeping at this time, the scores will be recorded when awake. Prior to discharge home, parents will be educated on use of the 0-10 pain scale and given a diary to keep an accurate record of postoperative pain issues through the study period. The goal is to capture maximum pain scores at rest and with movement. Patient and parental satisfaction with pain management and with the global perioperative experience will also be graded on a numeric scale 0-10 scale.

Time to readiness for discharge will also be measured from the time the patient enters the PACU to when the patient attains an Aldrete score of 9-10. This is a standardized scale used to assess discharge readiness at TCH and is listed below:

Aldrete Scoring System Activity Can move voluntarily or on command 4 extremities 2 2 extremities 1 0 extremities 0 Respiration Can deep-breathe and cough freely 2 Dyspnea, shallow or limited breathing 1 Apneic 0 Circulation Preoperative BP (mmHg) BP ± 20 mmHg of baseline 2 BP ± 20-50 mmHg of baseline 1 BP ± 20 mmHg 0 Consciousness Fully Awake 2 Arousable on calling 1 Not responding 0 Color Normal 2 Pale, dusky, blotchy 1 Cyanotic 0 Score of 10: ready for discharge

If the patient is discharged before the end of a 48 hour period after surgery, they will be given a diary to complete to list all medications given, and to assess their pain at various time intervals (12,24, 48 hours after surgery), along with their satisfaction with pain control. The patient will be contacted after discharge to obtain the data in the diary. Phone calls will also be placed on Post- operative Day (POD) #1,2, & 3 to the family following to assess measured endpoints (pain, medication usage, satisfaction, resolution of nerve block).

At the time of their follow up visit to the surgeon, a complete physical examination will be done including a neurological evaluation for any nerve injury.

ELIGIBILITY:
Inclusion Criteria:

1) Supracondylar fracture (2) Age 2-17 years (3) American Society of Anesthesiologists Status 1 -3 (4) Scheduled for closed reduction with percutaneous pinning under general anesthesia

Exclusion Criteria:

1. Pulseless extremity
2. Compromised neurologic status on exam (specifically assessment of radial, ulnar, and median nerve)
3. Known allergy to local anesthetics (7) Not scheduled for closed reduction with percutaneous pinning under general anesthesia
4. Bleeding diathesis
5. American Society of Anesthesiologist (ASA) status 4 or higher.
6. Sleep apnea by polysomnography

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2011-03-10 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Glover, MD, Principal Investigator — Baylor College of Medicine; Melissa Challman, MPH, Study Director — Baylor College of Medicine
Locations (1):
- Texas Children't Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: In-Hospital Data
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids
Started (Randomized) | 40 | 38
Completed | 35 | 38
Not Completed | 5 | 0
Not completed — Surgery cancelled | 1 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Physician Decision | 1 | 0
Period: 48-Hour Post-Discharge Data
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids
Started | 35 | 38
Completed | 21 | 18
Not Completed | 14 | 20
Not completed — Did not return diary | 14 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids | Total
Number analyzed (Participants) | 35 | 38 | 73
Age, Continuous [Median (Full Range); unit: years] | 6.52 [4.21 to 11.39] | 6.01 [3.84 to 10.2] | 6.09 [3.84 to 11.39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 20 | 21 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 35 | 38 | 73
ASA Physical Status [Count of Participants; unit: Participants] — The ASA Physical Status Classification System assesses and communicates a patient's pre-anesthesia medical co-morbidities. The ASA System ranges from I to VI with lower scores indicating healthy patients with no systemic disease. ASA I is a normal healthy patient and an ASA VI is a declared brain-dead patient whose organs are being removed for donor purposes.
  Participants
    ASA I | 25 | 27 | 52
    ASA II | 10 | 11 | 21
Weight [Mean (Standard Deviation); unit: kg] | 24.89 (8.07) | 23.75 (5.43) | 24.29 (6.85)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Opioid administration measured in mg/kg. Results below represent the total opioids given in the PACU, after discharge from the PACU, and then total post-operative period.
Time Frame: up to 48 hours after surgery
Population: Total PACU consumption was able to be calculated for all subjects. Not every subject returned their 48-hour diary. As such, the discharge consumption does not reflect all possible subjects.
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids
Number analyzed (Participants) | 35 | 38
mg/kg
  Total Intraoperative Opioids | 0 [0 to 0.09] | 0.2 [0.11 to 0.26]
  PACU - 1st 2 hours | 0 [0 to 0.05] | 0.12 [0.06 to 0.22]
  Home - Hour 2 to 48: number analyzed (Participants) | 22 | 19
  Home - Hour 2 to 48 | 0.25 [0 to 0.53] | 0.04 [0 to 0.53]
  Total Opioid Consumption - PACU and Home | 0.31 [0.05 to 0.53] | 0.26 [0.10 to 0.58]

2. Secondary Outcome: Time of First Analgesia Request
Description: Time at which additional analgesia was requested and/or administered by the nurse while in the PACU. Discharge data not reported due to poor diary return compliance.
Time Frame: PACU Period up to 3 hours
Population: Reflects only subjects who requested analgesia in the PACU.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids
Number analyzed (Participants) | 9 | 35
Minutes | 76 [53 to 93] | 27 [13 to 43]

3. Secondary Outcome: Time of Achieving Discharge Readiness
Description: Documented time that patient achieves an Aldrete Score of 9 -10. This is a standardized scale used to assess discharge readiness at Texas Children's Hospital.
Time Frame: From the time of PACU arrival up to time the patient achieves an Aldrete Score of 9- 10.
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids
Number analyzed (Participants) | 35 | 38
Minutes | 72 [30 to 125] | 94 [48 to 187]

4. Secondary Outcome: Incidence of Side Effects
Description: Documented side effects such as nausea, vomiting, pruritus, and respiratory depression.
Time Frame: up to 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids
Number analyzed (Participants) | 35 | 38
Participants
  Nausea | 1 | 0
  Vomiting | 0 | 0
  Pruritus | 0 | 0
  Respiratory Depression | 2 | 0

5. Secondary Outcome: Patient and Parent Satisfaction
Description: Child subject and parent satisfaction with pain management was measured using the global perioperative experience graded on a numeric scale of 0 - 10, with 0 indicating poor management to 10 indicating excellent pain management. Satisfaction is reported at 12-, 24-, 48-hours, and overall at home.
Time Frame: up to 48 hours after surgery
Population: Not all subjects returned their 48-hour diary.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids
Number analyzed (Participants) | 19 | 17
units on a scale
  Child's Satisfaction - at 12-hours: number analyzed (Participants) | 17 | 16
  Child's Satisfaction - at 12-hours | 5.8 [0 to 10] | 6.6 [0 to 10]
  Child's Satisfaction - at 24-hours: number analyzed (Participants) | 17 | 15
  Child's Satisfaction - at 24-hours | 5.6 [0 to 10] | 5.6 [0 to 10]
  Child's Satisfaction - at 48-hours: number analyzed (Participants) | 15 | 13
  Child's Satisfaction - at 48-hours | 7.5 [0 to 10] | 7.1 [0 to 10]
  Child's Satisfaction - Total time at home: number analyzed (Participants) | 18 | 16
  Child's Satisfaction - Total time at home | 6.1 [0 to 10] | 5.9 [0 to 10]
  Parent's Satisfaction - at 12-hours: number analyzed (Participants) | 18 | 17
  Parent's Satisfaction - at 12-hours | 5.8 [0 to 10] | 7.1 [0 to 10]
  Parent's Satisfaction - at 24-hours: number analyzed (Participants) | 18 | 16
  Parent's Satisfaction - at 24-hours | 6.4 [0 to 10] | 6.5 [0 to 10]
  Parent's Satisfaction - at 48-hours: number analyzed (Participants) | 17 | 14
  Parent's Satisfaction - at 48-hours | 8.1 [0 to 10] | 7.6 [0 to 10]
  Parent's Satisfaction - Total time at home | 7.9 [0 to 10] | 6.5 [0 to 10]

6. Secondary Outcome: The Mean Pain Score in the Postoperative Period
Description: The Verbal Numeric Scale (VNS) asks patients to verbally state a number between 0 and 10 that corresponds to their present pain intensity. 0 = no pain and 10 = worst possible pain ever. Pain was measured by the child subject in the PACU at arrival, 15-, 30-, 60- and 120-minutes. Pain was assessed by the child subject and a parent at home at 12-, 24-, and 48-hours after surgery. The results represent a mean of all verbal pain scores in the PACU, while at home, and overall.
Time Frame: From admission to PACU to 48 hours after surgery
Population: Some subjects in the PACU did not have VNS collected. In addition, not all of the 48-hour diaries were returned to allow for at home calculations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids
Number analyzed (Participants) | 35 | 38
units on a scale
  PACU: number analyzed (Participants) | 30 | 33
  PACU | 1.28 (1.88) | 4.76 (2.84)
  Home: number analyzed (Participants) | 19 | 17
  Home | 3.85 (2.55) | 3.49 (2.63)
  PACU + Home: number analyzed (Participants) | 31 | 34
  PACU + Home | 2.46 (2.44) | 4.44 (2.72)

ADVERSE EVENTS:
Time Frame: up to 48 hours after surgery
Arm/Group | Ultrasound Guided Supraclavicular Block | IV Opioids
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/38
Other Adverse Events (participants affected / at risk) | 0/35 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT02056288/Prot_SAP_000.pdf